CLINICAL TRIAL: NCT06779812
Title: Impact of Auriculotherapy on Postoperative Pain in Patients Undergoing Surgery for SCC. Parallel, Randomized, and Double-Blind Comparative Study
Brief Title: Impact of Auriculotherapy on Postoperative Pain in Patients Undergoing Surgery for SCC
Acronym: AURDO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Bizet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024-A02150-47
Record Dates: First submitted 2025-01-08; First posted 2025-01-17 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Pain After Carpal Tunnel Surgery

STUDY DESIGN:
Intervention Model Description: Group A (Experimental): Real auriculotherapy + standard medical care Group B (Control): Sham auriculotherapy + standard medical care
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Real auriculotherapy + standard medical care
  Interventions: Procedure: Carpal Tunnel Surgery; Other: real auricolothery
- Group B (Sham Comparator): Sham auriculotherapy + standard medical care
  Interventions: Procedure: Carpal Tunnel Surgery; Other: sham auriculotherapy

INTERVENTIONS:
Procedure: Carpal Tunnel Surgery — Carpal tunnel surgery is performed endoscopically, using smaller incisions. Endoscopic surgery is a minimally invasive method that allows for faster and less painful recovery
Other: real auricolothery — 3 days before the intervention, patients will have an auriculotherapy session with an experimental group
  Arms: Group A
Other: sham auriculotherapy — 3 days before the intervention, patients will have an auriculotherapy session with an sham group
  Arms: Group B

SUMMARY:
Auriculotherapy shows promising potential for pain management in patients with carpal tunnel syndrome (CTS). Studies have demonstrated encouraging results in pain reduction and improvement in quality of life. However, further research is required to strengthen these findings and fully integrate auriculotherapy into standard treatment protocols for CTS.

this prospective, double-blind comparative study aims to evaluate the effectiveness of auricular acupuncture in managing postoperative pain following outpatient carpal tunnel surgery

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged over 20 years
* Patients with carpal tunnel syndrome scheduled for endoscopic surgery
* Patients who have never undergone auriculotherapy sessions before
* No participation in another clinical study

Exclusion Criteria:

* Patients under 20 years of age
* Unable to undergo medical follow-up for the study
* Legally protected adult subjects, under guardianship or curatorship

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Postoperative Pain After Carpal Tunnel Surgery From Day 1 to Day 3, Based on Real or Sham Auriculotherapy Sessions | day1 to day 3
  Visual analog scale

SECONDARY OUTCOMES:
Evaluation of the Effects of Real or Sham Auriculotherapy Sessions on Analgesic Consumption | Follow-up Logbook from Day 1 to Day 3
  Analgesic Consumption

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Benkessou, Paris
  - Bizet Clinic, Paris

IPD SHARING:
Plan to Share IPD: Undecided